CLINICAL TRIAL: NCT04368845
Title: A Telerehabilitation Approach to Improve Long-term Physical Ability and Quality of Life in Patients With Severe Acute Respiratory Syndrome Coronavirus (SARSCoV-2, COVID-19) Immediately After Hospitalization. The ATHLOS Study
Brief Title: Telerehabilitation in Patients With COVID-19 After Hospitalization. The ATHLOS Study
Acronym: ATHLOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: University of Athens (Other); University of Ioannina (Other)
Responsible Party: Principal Investigator, Eleni Kortianou, Associate Professor in Respiratory Physiotherapy, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2020-04-20; First posted 2020-04-30 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2022-01

CONDITIONS: COVID-19; Comorbidities and Coexisting Conditions
Keywords: covid-19; telerehabilitation; physiotherapy; home rehabilitation
MeSH Terms: conditions — COVID-19 | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Two arm single blinded randomized control trial
Who Masked: Outcomes Assessor
Masking Description: Block Randomisation, Initial and final outcome assessors blinded to treatment arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Intervention Arm: Telerehabilitation (Active Comparator): The treatment arm will be given up to 1-hour resistive training exercises, breathing exercises and aerobic exercises administered by an expert physiotherapist via teleconference (telerehabilitation). Every ten days one physiotherapist will record the individualized exercise program, will reevaluate the magnitude of exercise for each patient and reinforce to continue or increase exercise magnitude.
  Interventions: Device: Telerehabilitation
- No Intervention: Conventional teleconference (No Intervention): The usual care arm will receive standard communication via teleconference every ten days for a six-month period without any specific recommendations and exercise prescription for home training. The control arm will be subject to the same assessments as the experimental arm at the start, and at the 3 and 6 months period.

INTERVENTIONS:
Device: Telerehabilitation — The treatment arm will be given up to 1-hour breathing exercises, aerobic and resistive training exercises administered by a physiotherapist via a telerehabilitation device every 10 days for a six-month period.
  Arms: Experimental Intervention Arm: Telerehabilitation

SUMMARY:
This is a two-phase multicenter study that will be conducted in collaboration with five university hospitals, in order to offer telehealth services at home in patients with COVID-19, after hospital discharge.

At the first phase an observational study aims to investigate the physical and psychological status of patients after hospital discharge and to provide support and information how to cope with symptoms (early fatigue, muscle weakness, eating difficulties, etc).

At the second phase a randomized control trial study will evaluate a 6-month telerehabilitation program for 100 adults (aged 20-65 years) diagnosed with COVID-19, who completed the first phase of this study. At this phase, the study will randomize (1:1 allocation) 100 male and female who were hospitalized with COVID-19 to either a 24-week home-based telerehabilitation program versus usual care. The intervention program includes individualized prescribed endurance exercises, low intensity aerobic exercises, upper and lower extremity strength training, breathing exercises as well as a three times per month online support with 1:1 supervision via video conferencing with an expert physiotherapist.

DETAILED DESCRIPTION:
This is a two-phase multicenter study that will be conducted in collaboration with five university hospitals in order to offer home telehealth services in patients with COVID-19, after hospital discharge.

At the first phase, an observational study aims to investigate the physical and psychological status of patients after hospital discharge and to provide support and information how to cope with symptoms (early fatigue, muscle weakness, eating difficulties, etc).

We aim to support 200 patients with age 20-65 years, between a 1-8 week period after hospital discharge, providing an e-book with body exercises, breathing exercises and nutritional support, additionally to four telehealth consultation sessions.

At the second phase, a single blinded randomized control trial study will evaluate a 6-month home telerehabilitation program for 100 diagnosed with COVID-19 adults (aged 20-65 years), who completed the first phase of this study. The second phase will randomize (1:1 allocation) 100 male and female who were hospitalized with COVID-19 to either a 24-week home-based telerehabilitation program versus usual care.

The intervention includes individualized prescribed upper and lower extremity endurance exercises, aerobic exercises, upper and lower extremity strength training, breathing exercises as well as a three times per month online support with 1:1 supervision via video conferencing with an expert physiotherapist.

The usual care group will be advised to follow the instructions of the e-book for any possible exercise training. Three times per month with 1:1 video conferencing, an expert physiotherapist will record any possible exercise with no further recommendations or support.

Changes from baseline in physical activity levels, cardiorespiratory fitness, physical performance, lower limb strength, anxiety and depression and health-related quality of life will be assessed at 3 and 6 months for both groups. All functional tests in the second phase of the study will be performed via supervision teleconference for all the participants with an expert physiotherapist. Findings from this project will contribute to the field of telerehabilitation in patients with COVID-19 after hospital discharge and will provide critical preliminary data for the design and implementation of a larger, randomized control trial assessing the impact of telerehabilitation on long-term clinical outcomes following infection or re-infection from coronaviruses.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults with age from 20 to 65 years hospitalized due COVID-19 infection. Able to give consent

Exclusion Criteria:

* the presence of mental illness, any physical disability that makes difficult to mobilize patients, severe heart disease, severe musculoskeletal pain, vascular aneurysms, severe neurological condition, pregnancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Physical Performance | Change From Baseline in SPPB Scores at 3 and 6 months
  The Short Physical Performance Battery (SPPB) is comprised of 3 tasks: a standing balance test (side by side, semi-tandem and tandem), a 4-m habitual gait speed, and 5 sit to stand from a chair. Each task is scored (based on time) from 0-4 points. The total score is 12 points and this represents the highest performance. It can be easily performed at home via video conferencing
Cardiorespiratory fitness | Change From Baseline in 3MST Scores at 3 and 6 months
  The 3 minute step test (3MST) is a field test designed to measure aerobic (cardiovascular) fitness. Participants step up and down a 30-cm high step for 3 minutes at a pace of 24 steps per minute. Oxygen saturation, heart rate and fatigue (using the Borg 0-10 scale) will be assessed at the beginning, at the end and every minute after full recovery in order to evaluate the heart's, fatigue and saturation recovery rates. Because it is a submaximal test it can easily be completed at home and administrated via video conferencing.
Lower limb Strength | Change From Baseline in STST Scores at 3 and 6 months
  The 30 sec sit-to-stand test (STST) is a feasible alternative for measuring lower limb muscle strength and endurance. The outcome is the number of times that the participant is able to completely stand up from the chair within 30 seconds.
Health Related Quality of Life | Change From Baseline in SF-36 Scores at 3 and 6 months
  The Short Form Health Survey (SF-36) consists of 36 questions spanning 8 health (physical and mental) domains. The eight domains are: vitality, physical functioning, bodily pain, general health, physical role functioning, emotional role functioning, social role and mental health. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. Converging the individual scores into z-score, a standardized score (mean 50) is provided for each domain allowing comparisons between populations. The lower the score the more disability. It is a valid patient-reported survey of health-related quality of life in patient populations and it is responsive to change following therapeutic interventions.
Anxiety and Depression | Change From Baseline in HADS Scores at 3 and 6 months
  Hospital anxiety and depression scale (HADS) is a 14-item questionnaire for screening anxiety (7 items) and depression (7 items). Each item is scored from 0-3 (a 4-point severity scale). Highest anxiety or depression score is 21. Patients are defined as having anxiety or depression or both if the score is 8 or more in the each subscale
Physical Activity | Change From Baseline in IPAQ Scores at 3 and 6 months
  The International Physical Activity Questionnaire (IPAQ) is a frequently used instrument for the evaluation of physical activity (PA). It was developed in order to assess physical activity in adults aged 18-65 years. The greek version of IPAQ, (IPAQ-Gr) sums up moderate, vigorous, walking physical activities over the previous seven-day period and generate a total physical activity score (PAscore), expressed in MET-minutes per week (MET.min.wk-1 ).
  Based on the IPAQ scoring procedure, physical activity status is classified into three categories (PAclasses): (1) low PAclass, insufficiently active subjects (total PAscore < 600 MET.min.wk-1); (2) moderate PAclass (total PAscore ≥ 600 MET.min.wk-1 or vigorous PAscore ≥ 480 MET.min.wk-1) and (3) high PAclass (total PAscore ≥ 3000 MET.min.wk-1 or vigorous PAscore ≥ 1500 MET.min.wk-1).

SECONDARY OUTCOMES:
Fatigue | Change From Baseline in Borg CR-10 Scores at 3 and 6 months
  The Borg CR-10 (CR= scale range) scale is a rating scale for self-reported dyspnea. 0 represents no symptoms and 10 the worst previously experienced symptoms.
Dyspnea | Change From Baseline in MMRC Scores at 3 and 6 months
  The modified Medical Research Council Dyspnea Scale (MMRC). A score from 0-4 is used to classify the impact of dyspnea on physical function in patients with respiratory limitations. 0 represents a person who suffers from dyspnea only with strenuous exercise. 4 represents a person who are to breathless to leave the house, or breathless when dressing/undressing.

CONTACTS AND LOCATIONS:
Overall Officials: ELENI KORTIANOU, PhD, PT, Study Director — Clinical Exercise Physiology and Rehabilitation Research Laboratory; ELENI KAPRELI, PhD, PT, Study Chair — Clinical Exercise Physiology and Rehabilitation Research Laboratory
Locations (1):
- Clinical exercise Physiology and rehabilitation research laboratory, Lamia, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papathanasiou G, Georgoudis G, Papandreou M, Spyropoulos P, Georgakopoulos D, Kalfakakou V, Evangelou A. Reliability measures of the short International Physical Activity Questionnaire (IPAQ) in Greek young adults. Hellenic J Cardiol. 2009 Jul-Aug;50(4):283-94. PMID 19622498
- [Background] Bergland A, Strand BH. Norwegian reference values for the Short Physical Performance Battery (SPPB): the Tromso Study. BMC Geriatr. 2019 Aug 8;19(1):216. doi: 10.1186/s12877-019-1234-8. PMID 31395008
- [Background] Wassenberg MW, Severs D, Bonten MJ. Psychological impact of short-term isolation measures in hospitalised patients. J Hosp Infect. 2010 Jun;75(2):124-7. doi: 10.1016/j.jhin.2010.01.023. Epub 2010 Apr 10. PMID 20381912